CLINICAL TRIAL: NCT05493423
Title: Confirmatory Study to Assess the V Needle in End-Stage Renal Disease Patients During In-Clinic Hemodialysis: Clinic-SAVER
Brief Title: Confirmatory Study to Assess the V Needle in End-Stage Renal Disease Patients During In-Clinic Hemodialysis
Acronym: Clinic-SAVER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hemotek Medical Inc (Industry)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CIP 001; 5R44DK101253 (NIH)
Record Dates: First submitted 2022-08-03; First posted 2022-08-09 (Actual); Results first posted 2025-02-05 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-01

CONDITIONS: End Stage Renal Disease
Keywords: hemodialysis; dialysis; dislodgement; venous needle; venous needle dislodgement; AV fistula set
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Needles

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Standard of Care vs. V Needle Performance Assessment (Experimental): Subjects will undergo three dialysis sessions using standard of care needles (control) and results will be compare to 6 dialysis sessions using the V Needle (experimental).
  Interventions: Device: V Needle AV Fistula Set

INTERVENTIONS:
Device: V Needle AV Fistula Set — Hemotek Medical Inc. has developed the V Needle, a new AV fistula set for hemodialysis designed to reduce patient risk from exsanguination-related injury or death during therapy. In the event of complete dislodgement of the V Needle from the arm during use, the V Needle is designed to activate, creating high line pressure designed to generate an automated dialysis machine blood pump shut down.
  Other Names: V Needle

SUMMARY:
This study is a prospective, multi-center, single-arm study with subjects acting as their own control designed to confirm the safety, performance, and usability of the V Needle, a new safety needle for use during in-clinic hemodialysis that is designed to automatically generate a partial occlusion of the internal fluid path and trigger the hemodialysis machine to alarm and shut off if a complete dislodgement of the venous needle from the arm inadvertently occurs.

DETAILED DESCRIPTION:
In patients undergoing hemodialysis for the treatment of end-stage renal disease, Venous Needle Dislodgement (VND) is a rare, but potentially fatal situation in which the needle delivering a patient's blood back to the body after filtration by a dialysis machine becomes inadvertently disconnected from the patient. Hemotek Medical Inc. has developed the V Needle, a venous needle return that is designed to reduce patient risk from exsanguination-related injury or death. This clinical study will serve as a confirmatory study to gain FDA marketing clearance of the Hemotek V Needle system in the clinical setting. During this study, the ability of the V Needle to successfully deliver appropriate hemodialysis therapy per the facility's guidelines will be assessed. It will also be used to determine if the V Needle triggers false blood alarms under normal operating conditions. This study will also be used to demonstrate the V Needle meets effective usability criteria. Rates of adverse events and ability to complete the hemodialysis session will be compared to the rates recorded using commercially available devices during the hemodialysis sessions prior to the use of the Hemotek V Needle.

The study is an open-label, non-randomized, single arm, multi-center trial with subject's serving as their own control. For the first three (3) control sessions, subjects will undergo usual hemodialysis sessions with a commercially available device. For the remaining six (6) sessions, subjects will be cannulated with a V Needle in place of a usual venous line AV fistula set.

The hemodialysis sessions will be conducted in the clinic. Subjects will be observed by a clinician for the duration of each session. Clinicians will monitor the session for any abnormal disruptions, therapy interruptions, and/or adverse events, including hemolysis, due to V Needle presence. All machine blood alarms, therapy interruptions, and/or partial or complete needle dislodgements will be recorded and immediately corrected. A clinician will perform cannulation.

Cannulation site and surrounding tissue will be examined by the nurse and assessed for any locally induced trauma before and after treatment. A survey will be completed by the clinicians and patients to assess usability, comfort, and feelings of safety of the V Needle.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with end-stage renal disease receiving chronic hemodialysis in a clinical setting.
2. Subjects must be able to receive hemodialysis with the Hemotek 15-gauge, 1 inch length V Needle, with 12 inch tubing.
3. Age greater than or equal to 22 years old at screening.
4. Vascular access via a mature arteriovenous (AV) fistula or graft in the arm and determined to be adequate for a chronic hemodialysis therapy.
5. AV fistula has already been demonstrated to adequately permit one or more hemodialysis sessions.
6. Subject prescribed blood flow rates between 200 ml/min and 450 ml/min
7. In women with child-bearing potential, negative urine or serum pregnancy test at Screening.
8. Subject able to communicate effectively with investigative staff, competent and willing to give written informed consent, and able to comply with entire study procedures.
9. Hemoglobin ≥9 g/dL (consistent with KDOQI guidelines)
10. Normal platelet count (≥150,000 /mm3)
11. International Normalized Ratio (INR) ≤ 1.5

Exclusion Criteria:

1. Subjects receiving chronic hemodialysis with a vascular catheter.
2. Subjects with vascular access that is determined by the clinician to be unacceptable for a hemodialysis procedure.
3. Patients with a bleeding diathesis
4. Patients receiving anti-coagulants
5. Previous vascular access surgery (≤30 days from study entry) or planned access surgery
6. Known hypersensitivity to any imaging agents (e.g., contrast) that may be required during the study period
7. Patients with confirmed vasculitis
8. Vascular access infection or systemic active infection within 30 days of study entry
9. Life expectancy less than 12 months
10. Planned renal transplantation or planned conversion to peritoneal dialysis
11. Subjects with any condition determined by the investigator that precludes them from safely participating in the study.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2022-11-07 (Actual); Primary Completion 2023-07-10 (Actual); Study Completion 2023-07-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wesley Calhoun, MD, Principal Investigator — Davita Clinical Research; Tahira Alves, MD, Principal Investigator — Davita Clinical Research
Locations (1):
- Davita, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from patients receiving hemodialysis three times per week at one of two Davita dialysis clinics in San Antonio, TX. 15 subjects total were evaluated and each subject served as their own control. So 15 subjects each had three control sessions followed by six V Needle sessions..
Groups:
- Standard of Care (Control) First, Then V Needle (Experimental): 15 Subjects served as their own controls and had three dialysis sessions using standard of care needles (control) over one week. Sessions were sequential. Dialysis session flow rates for 11 of these patients was 400 mL/min and flow rate for 4 of these patients was 450 mL/min.
  The same 15 subjects then had six dialysis sessions over the next two weeks using the Hemotek V Needle (test article, experimental) at the same assigned flow rates. Sessions were sequential.
Period: Standard of Care (Control) 3x - One Week
Arm/Group | Standard of Care (Control) First, Then V Needle (Experimental)
Started | 15 (In this period, subjects are using the control device only for 3 sessions over one week)
400 mL/Min Flow Rate | 11
450 mL/Min Flow Rate | 4
Completed | 15
Not Completed | 0
Period: V Needle (Experimental) 6x - Two Weeks
Arm/Group | Standard of Care (Control) First, Then V Needle (Experimental)
Started | 15 (In this second period, subjects are using only the experimental device (the V Needle) for 6 sessions over two weeks.)
400 mL/Min Flow Rate | 11
450 mL/Min Flow Rate | 4
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All 15 subjects served as their own controls.
Groups:
- Standard of Care vs. V Needle Performance Assessment: Subjects serve as their own controls in this study. They will undergo three dialysis sessions using standard of care needles (control sessions) and those results will be compared to 6 dialysis sessions using the V Needle (test sessions). THEREFORE, WE DO NOT USE A "BASELINE MEASURE" HERE BUT INSTEAD INCLUDE A 'CONTROL ARM' IN THE OUTCOME MEASURES SECTIONS.
Arm/Group | Standard of Care vs. V Needle Performance Assessment
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.7 (10.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Information determined during enrollment interview
  Participants
    Hispanic or Latino | 10
    Not Hispanic or Latino | 5
    Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 1
  White | 13
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Successful Hemodialysis Sessions
Description: A successful hemodialysis session is one in which the physician's dialysis prescription has been appropriately delivered. There are only two options for results: successful or unsuccessful. Success rates will be calculated for 3 control sessions using standard of care needles and compared with the average success rate determined from 6 experimental V Needle sessions.
Time Frame: 3 weeks total: 1 week for 3 control sessions and 2 weeks for 6 experimental (V Needle) sessions per subject
Population: Study subjects who meet eligibility criteria at each site
Measure: Number; unit: percentage of successful sessions
Units Other Than Participants: Sessions
Groups:
- Control Device: All subjects using SysLoc Mini
- Test Device: All subjects using V Needle
Arm/Group | Control Device | Test Device
Number analyzed (Participants) | 15 | 15
Number analyzed (Sessions) | 45 | 90
percentage of successful sessions | 100 | 98.9
Statistical Analysis 1: Comparison: Control Device vs Test Device; Test type: Non-Inferiority — The null hypothesis is that the difference between the rates of completed hemodialysis sessions for the test and control groups is less than or equal to the non-inferiority margin (indicating inferior success rate). Rejection of the null hypothesis indicates the data supports the alternative hypothesis that the difference between the rates of successfully completed HD sessions for the test and control groups is at least the non-inferiority margin (indicating non-inferior success rate); p = .008, Farrington-Manning; non-inferiority margin = 0.08
Statistical Analysis 2: Comparison: Control Device vs Test Device; Test type: Equivalence — non-inferiority margin = 0.08; p = .002, Equivalence Test with paired data

2. Other Pre Specified Outcome: Machine Alarm Rate (Blood Alarms Only) During Hemodialysis Therapy Sessions, Including False Alarms.
Description: The hemodialysis machine alarm rate will be monitored per session and then averaged and compared for three control sessions using standard of care needles and then again for six experimental V Needle sessions.
Time Frame: 3 weeks total: 1 week for 3 control sessions and 2 weeks for 6 experimental (V Needle) sessions per subject
Population: The same 15 subjects served as their own controls.
Measure: Mean (Standard Deviation); unit: alarms/session
Units Other Than Participants: Sessions
Arm/Group | Control Device | Test Device
Number analyzed (Participants) | 15 | 15
Number analyzed (Sessions) | 45 | 90
alarms/session | 1.11 (0.25) | 1.92 (0.51)
Statistical Analysis 1: Comparison: Control Device vs Test Device; Test type: Superiority; p = 0, t-test, 2 sided — The p-value was calculated, but was low enough to be rounded down to 0 by the statistical software

3. Other Pre Specified Outcome: False Alarms Per Session (as a % of All Venous Alarms Per Same Session)
Description: Overall false alarm rate per hemodialysis session as determined as a percentage of all venous alarms.
Time Frame: 3 weeks (time required to complete all control and test dialysis sessions per patient)
Measure: Number; unit: percentage of false alarms
Units Other Than Participants: Venous Alarms
Groups:
- Standard of Care (Baseline/Control) Performance Assessment: Subjects will undergo three dialysis sessions using standard of care needles (control). Sessions are sequential and unless otherwise noted takes one week to complete three sessions. Flow rate for 11 of these patients was 400 mL/min and flow rate for 4 of these patients was 450 mL/min.
- V Needle (Test) Performance Assessment: Subjects will undergo six dialysis sessions using the Hemotek V Needle (test article). Sessions are sequential and unless otherwise noted takes two weeks to complete six sessions. Flow rate for these 11 patients was 400 mL/min and flow rate for 4 of these patients was 450 mL/min.
Arm/Group | Standard of Care (Baseline/Control) Performance Assessment | V Needle (Test) Performance Assessment
Number analyzed (Participants) | 15 | 15
Number analyzed (Venous Alarms) | 6 | 32
percentage of false alarms | 82 | 83.66
Statistical Analysis 1: Comparison: Standard of Care (Baseline/Control) Performance Assessment vs V Needle (Test) Performance Assessment; Test type: Superiority; p = 0.84, t-test, 2 sided — P < 0.05 is considered significant

4. Other Pre Specified Outcome: Venous Alarm Rate (All) Per Session
Description: Rate of venous alarms per hemodialysis session
Time Frame: 3 weeks total: 1 week for 3 control sessions and 2 weeks for 6 experimental (V Needle) sessions per subject
Measure: Mean (Standard Deviation); unit: venous alarms/session
Units Other Than Participants: Alarms
Arm/Group | Standard of Care (Baseline/Control) Performance Assessment | V Needle (Test) Performance Assessment
Number analyzed (Participants) | 15 | 15
Number analyzed (Alarms) | 45 | 90
venous alarms/session | 0.14 (0.43) | 0.36 (0.38)
Statistical Analysis 1: Comparison: Standard of Care (Baseline/Control) Performance Assessment vs V Needle (Test) Performance Assessment; Test type: Superiority; p = 0.132, t-test, 2 sided

5. Other Pre Specified Outcome: % All (False) Alarms Related to V Needle Footplate Opening Inappropriately
Description: % All (false) Alarms Related to V Needle footplate opening inappropriately during each hemodialysis session
Time Frame: 3 weeks total: 1 week for 3 control sessions and 2 weeks for 6 experimental (V Needle) sessions per subject
Population: There are 0 units analyzed in the control arm because the control device does not have a protective footplate to assess.
Measure: Number; unit: % All (false) Alarms Related to V Needle
Units Other Than Participants: Alarms
Arm/Group | Standard of Care (Baseline/Control) Performance Assessment | V Needle (Test) Performance Assessment
Number analyzed (Participants) | 15 | 15
Number analyzed (Alarms) | 0 | 13
% All (false) Alarms Related to V Needle |  | 0
Statistical Analysis 1: Comparison: Standard of Care (Baseline/Control) Performance Assessment vs V Needle (Test) Performance Assessment; Test type: Superiority; p = 0.84, t-test, 2 sided — P < 0.05 is considered significant

6. Other Pre Specified Outcome: % All Alarms Related to Venous Needle
Description: % of all alarms related to Venous needle per hemodialysis session
Time Frame: 3 weeks total: 1 week for 3 control sessions and 2 weeks for 6 experimental (V Needle) sessions per subject
Measure: Number; unit: % of all alarms related to venous needle
Units Other Than Participants: Alarms
Arm/Group | Standard of Care (Baseline/Control) Performance Assessment | V Needle (Test) Performance Assessment
Number analyzed (Participants) | 15 | 15
Number analyzed (Alarms) | 50 | 173
% of all alarms related to venous needle | 12 | 18
Statistical Analysis 1: Comparison: Standard of Care (Baseline/Control) Performance Assessment vs V Needle (Test) Performance Assessment; Test type: Superiority; p = 0.197, t-test, 2 sided — P < 0.05 is considered significant

7. Other Pre Specified Outcome: % Hemodialysis Sessions Requiring a Change to Blood Flow Rate Setting During Therapy
Description: Percentage of the hemodialyis sessions during which the clinical staff was required to change the original blood flow rate setting during therapy sessions
Time Frame: 3 weeks total: 1 week for 3 control sessions and 2 weeks for 6 experimental (V Needle) sessions per subject
Measure: Number; unit: percentage of hemodialysis sessions
Units Other Than Participants: Sessions
Arm/Group | Standard of Care (Baseline/Control) Performance Assessment | V Needle (Test) Performance Assessment
Number analyzed (Participants) | 15 | 15
Number analyzed (Sessions) | 45 | 90
percentage of hemodialysis sessions | 6.67 | 3.33
Statistical Analysis 1: Comparison: Standard of Care (Baseline/Control) Performance Assessment vs V Needle (Test) Performance Assessment; Test type: Superiority; p = 0.424, t-test, 2 sided

8. Other Pre Specified Outcome: Mean Venous Pressure (in mm Hg) Per Hemodialyis Session for Subjects Dialyzing at 400 mL/Min
Description: Mean Venous Pressure (in mm Hg) per hemodialysis session for subjects dialyzing at a flow rate of 400 mL/min
Time Frame: 3 weeks total: 1 week for 3 control sessions and 2 weeks for 6 experimental (V Needle) sessions per subject
Measure: Mean (Standard Deviation); unit: mm Hg/session
Units Other Than Participants: Sessions
Arm/Group | Standard of Care (Baseline/Control) Performance Assessment | V Needle (Test) Performance Assessment
Number analyzed (Participants) | 11 | 11
Number analyzed (Sessions) | 33 | 66
mm Hg/session | 179 (31) | 208 (37)
Statistical Analysis 1: Comparison: Standard of Care (Baseline/Control) Performance Assessment vs V Needle (Test) Performance Assessment; Test type: Superiority; p = 0, t-test, 2 sided — The p-value was calculated, but was low enough to be rounded down to 0 by the statistical software

9. Other Pre Specified Outcome: Mean Venous Pressure (in mm Hg) Per Hemodialyis Session for Subjects Dialyzing at 450 mL/Min
Description: Mean Venous Pressure (in mm Hg_) per hemodialysis session for subjects dialyzing at a flow rate of 450 mL/min
Time Frame: 3 weeks total: 1 week for 3 control sessions and 2 weeks for 6 experimental (V Needle) sessions per subject
Measure: Mean (Standard Deviation); unit: mm Hg/session
Units Other Than Participants: Sessions
Arm/Group | Standard of Care (Baseline/Control) Performance Assessment | V Needle (Test) Performance Assessment
Number analyzed (Participants) | 4 | 4
Number analyzed (Sessions) | 12 | 24
mm Hg/session | 213 (30) | 247 (35)
Statistical Analysis 1: Comparison: Standard of Care (Baseline/Control) Performance Assessment vs V Needle (Test) Performance Assessment; Test type: Superiority; p = 0, t-test, 2 sided — The p-value was calculated, but was low enough to be rounded down to as 0 by the statistical software

10. Other Pre Specified Outcome: Mean Transmembrane Pressure (in mm Hg) Per Session for Subjects Dialyzing at 400 mL/Min
Description: Mean Transmembrane Pressure (mm Hg) per hemodialysis session for subjects dialyzing at 400 mL/min
Time Frame: 3 weeks total: 1 week for 3 control sessions and 2 weeks for 6 experimental (V Needle) sessions per subject
Measure: Mean (Standard Deviation); unit: mm Hg/session
Units Other Than Participants: Sessions
Arm/Group | Standard of Care (Baseline/Control) Performance Assessment | V Needle (Test) Performance Assessment
Number analyzed (Participants) | 11 | 11
Number analyzed (Sessions) | 33 | 66
mm Hg/session | 48 (17) | 48 (16)
Statistical Analysis 1: Comparison: Standard of Care (Baseline/Control) Performance Assessment vs V Needle (Test) Performance Assessment; Test type: Superiority; p = 0.57, t-test, 2 sided — P < 0.05 is considered significant

11. Other Pre Specified Outcome: Mean Transmembrane Pressure (mm Hg) Per Session for Subjects Dialyzing at 450 mL/Min
Description: Mean Transmembrane Pressure (mm Hg) per hemodialysis session for subjects dialyzing at 450 mL/min
Time Frame: 3 weeks total: 1 week for 3 control sessions and 2 weeks for 6 experimental (V Needle) sessions per subject
Measure: Mean (Standard Deviation); unit: mm Hg/session
Units Other Than Participants: Sessions
Arm/Group | Standard of Care (Baseline/Control) Performance Assessment | V Needle (Test) Performance Assessment
Number analyzed (Participants) | 4 | 4
Number analyzed (Sessions) | 12 | 24
mm Hg/session | 43 (14) | 44 (13)
Statistical Analysis 1: Comparison: Standard of Care (Baseline/Control) Performance Assessment vs V Needle (Test) Performance Assessment; Test type: Superiority; p = 0, t-test, 2 sided — The p-value was calculated, but was low enough to be rounded down to 0 by the statistical software

12. Other Pre Specified Outcome: Mean Arterial Pressure (in mm Hg) Per Session for Subjects Dialyzing at a Flow Rate 400 mL/Min
Description: Mean Arterial Pressure (mm Hg) per each session for subjects dialyzing at a flow rate of 400 mL/min
Time Frame: 3 weeks total: 1 week for 3 control sessions and 2 weeks for 6 experimental (V Needle) sessions per subject
Measure: Mean (Standard Deviation); unit: mm Hg/session
Units Other Than Participants: Sessions
Arm/Group | Standard of Care (Baseline/Control) Performance Assessment | V Needle (Test) Performance Assessment
Number analyzed (Participants) | 11 | 11
Number analyzed (Sessions) | 33 | 66
mm Hg/session | -167 (32) | -175 (36)
Statistical Analysis 1: Comparison: Standard of Care (Baseline/Control) Performance Assessment vs V Needle (Test) Performance Assessment; Test type: Superiority; p = 0.211, t-test, 2 sided

13. Other Pre Specified Outcome: Mean Arterial Pressure (in mm Hg) Per Session for Subjects Dialyzing at a Flow Rate 450 mL/Min
Description: Mean Arterial Pressure (mm Hg) per session for those subjects dialyzing at a flow rate of 450 mL/min
Time Frame: 3 weeks total: 1 week for 3 control sessions and 2 weeks for 6 experimental (V Needle) sessions per subject
Measure: Mean (Standard Deviation); unit: mm Hg/session
Units Other Than Participants: Sessions
Arm/Group | Standard of Care (Baseline/Control) Performance Assessment | V Needle (Test) Performance Assessment
Number analyzed (Participants) | 4 | 4
Number analyzed (Sessions) | 12 | 24
mm Hg/session | -197 (37) | -199 (29)
Statistical Analysis 1: Comparison: Standard of Care (Baseline/Control) Performance Assessment vs V Needle (Test) Performance Assessment; Test type: Superiority; p = 0.804, t-test, 2 sided — P < 0.05 is considered significant

14. Other Pre Specified Outcome: % Hemodialysis Sessions Where 'Achieved' Blood Flow Rate is Within 75% of 'Prescribed' Blood Flow Rate
Description: Variations of the blood flow rate will be monitored to determine if the achieved blood flow rate during a given session is within 75% of the prescribed blood flow rate. Assessments will be determined for three control sessions using standard of care needles and for six V Needle sessions.
Time Frame: 3 weeks total: 1 week for 3 control sessions and 2 weeks for 6 experimental (V Needle) sessions per subject
Population: Study subjects who meet eligibility criteria at each site
Measure: Number; unit: percentage of sessions
Units Other Than Participants: Sessions
Arm/Group | Control Device | Test Device
Number analyzed (Participants) | 15 | 15
Number analyzed (Sessions) | 45 | 90
percentage of sessions | 95.6 | 98.9
Statistical Analysis 1: Comparison: Control Device vs Test Device; Test type: Superiority; p = 0.307, t-test, 2 sided — P < 0.05 is considered significant

15. Other Pre Specified Outcome: % Sessions Where Clinician Was Able to Successfully Cannulate Fistula
Description: The clinician will self-report if the fistula was successfully cannulated (a yes or no metric) for three control sessions using standard of care needles and for six V Needle test sessions.
Time Frame: 3 weeks total: 1 week for 3 control sessions and 2 weeks for 6 experimental (V Needle) sessions per subject
Population: Study subjects who meet eligibility criteria at each site
Measure: Number; unit: percentage of hemodialysis sessions
Units Other Than Participants: Sessions
Arm/Group | Control Device | Test Device
Number analyzed (Participants) | 15 | 15
Number analyzed (Sessions) | 45 | 90
percentage of hemodialysis sessions | 100 | 98.9
Statistical Analysis 1: Comparison: Control Device vs Test Device; Test type: Superiority; p = 0.315, t-test, 2 sided — P < 0.05 is considered significant

ADVERSE EVENTS:
Time Frame: All AE data and outcomes data was captured per session, with 3 control sessions, in the first week, followed by 6 experimental sessions over the next two weeks, resulting in a three week data collection period per subject. Additionally, all subjects were followed for 7 more days following each of their study dialysis sessions to observe for any potential AEs. Thus, data collection coupled with AE observation resulted in an overall observation period of 4 weeks total per subject.
Description: Patients were monitored during and after therapy for the appearance of any AE's or potential symptoms of AE's. Patient medical records were tracked between each session. Follow-up contact was made 7 days following the last study session to determine if any AE's or potential symptoms of AE's had occurred. Patients had clinical study coordinator contact information to self-report any other potential AE's or potential symptoms of AE's.
Groups:
- Control Device: All subjects using SysLoc Mini, the Standard of Care (control).
- Test Device: All subjects using V Needle, the test device (experimental). These subjects are the same as the control arm.
Arm/Group | Control Device | Test Device
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 1/15
Other Adverse Events (participants affected / at risk) | 1/15 | 2/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control Device (N=15) | Test Device (N=15)
High Blood Pressure (General disorders) | 0 (0) | 1 (1)
Lung Edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control Device (N=15) | Test Device (N=15)
SYNCOPE (Vascular disorders) | 1 (1) | 0 (0)
CLOT (Vascular disorders) | 0 (0) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-04-10): https://cdn.clinicaltrials.gov/large-docs/23/NCT05493423/Prot_SAP_001.pdf